CLINICAL TRIAL: NCT03210220
Title: Efficacy of Preoperative Ultrasound Guided Pectoral Nerve Block for Intraoperative Opioid Sparing Effect and Postoperative Analgesia in Patients Undergoing Surgery for Breast Cancer.
Brief Title: Efficacy of Preoperative Pectoral Nerve Block for Intraoperative Opioid Sparing Effect and Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Jung Ju Choi, assistance professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: PENBreast
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients either received the Pecs II block (Pecs group) or did not receive it (control group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One anesthesiologist (JJC) performed all blocks in the Pecs group enrolled patients. After the intervention, the participants and the investigator responsible for the study outcome assessment were blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pecs group (Experimental): Ultrasound guided pectoral nerve block is performed right after induction, before surgery. The needle is advanced to the tissue plane between the pectoralis major and pectoralis minor muscle at the vicinity of the pectoral branch of the acromiothoracic artery, and 10 mL of 0.5% ropivacaine deposited. In a similar manner, 20 mL is deposited at the level of the third rib between the pectoralis minor muscle and the serratus anterior muscle .
  Interventions: Procedure: Pecs II block
- control group (No Intervention): There is no block.

INTERVENTIONS:
Procedure: Pecs II block — After identifying the axillary vein and artery, the ultrasound probe was positioned inferio-laterally, between the 3rd and 4th ribs, and then the pectoralis major and minor, and serratus anterior muscles were confirmed. The needle was advanced in a medio-lateral direction in-plane view of the ultrasound. For the Pecs II block, a total 30 mL of 0.5% ropivacaine was injected. First, the needle tip was advanced into the fascia between the pectoralis major and minor muscles and 10 mL of 0.5% ropivacaine was injected. Thereafter, the needle tip was advanced into the tissue plane between the pectoralis minor and serratus anterior muscles, and 20 mL of 0.5% ropivacaine was injected in a similar manner.
  Arms: pecs group

SUMMARY:
The purpose of this study is to determine whether pectoral nerves blocks（PECS） would reduces the opioid consumption during the surgery and postoperative pain after breast cancer surgery.

DETAILED DESCRIPTION:
Forty adult female participants scheduled for elective breast cancer surgery under general anesthesia are randomly allocated to receive either general anesthesia plus Pecs block(Pecs group, n=20) or general anesthesia alone (control group, n=20).

After arrived in the operating room，all patients undergo operation under total intravenous anesthesia (TIVA) with or without pectoral nerves blocks(PECS) . After anesthesia induction，the participants in the Pecs group receive an ultrasound-guided Pecs block before the start of the operation.

Pecs block technology：After cleaning the infraclavicular and axillary regions , the linear probe is placed below the lateral third of the clavicle. After recognition of the appropriate anatomical structures, then the block is performed . The needle is advanced to the tissue plane between the pectoralis major and pectoralis minor muscle at the vicinity of the pectoral branch of the acromiothoracic artery, and 10 mL of 0.5% ropivacaine deposited. In a similar manner, 20 mL is deposited at the level of the third rib between the pectoralis minor muscle and the serratus anterior muscle .

During operation the remifentanil administration in each group is guided using the surgical pleth index( SPI). the SPI target range was 20 to 50 Anesthetic depth is maintained and continuously adjusted with propofol to achieve Bispectral Index (BIS) between 40 and 60.

primary outcome intraoperative remifentanil consumption secondaty outcome postoperative pain score and rescue analgesic requirement

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists( ASA) I or II Scheduled for breast cancer surgery

Exclusion Criteria:

Sensitivity to local anesthetic, Bleeding disorders , Receiving anticoagulant, Body mass index (BMI) > 35/kg/m2 , Spine or chest wall deformity , Pregnancy

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Cheon Lee, Study Chair — Gachon University Gil Medical Center
Locations (1):
- Kyung Cheon Lee, Incheon, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pecs Group | Control Group
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pecs Group | Control Group | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (7.71) | 52.7 (9.22) | 52.07 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 19 | 20 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 19 | 20 | 39
weight [Mean (Standard Deviation); unit: kg] | 59.4 (10) | 63.5 (8) | 61.5 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Remifentanil Consumption
Description: Intraoperative remifentanil consumption during surgery(whole intraoperative period)
Time Frame: whole intraoperative period
Measure: Mean (Standard Deviation); unit: μg/kg/h
Arm/Group | Pecs Group | Control Group
Number analyzed (Participants) | 19 | 20
μg/kg/h | 6.75 (2.18) | 10.12 (3.68)

ADVERSE EVENTS:
Time Frame: 3days
Arm/Group | Pecs Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03210220/Prot_SAP_000.pdf